CLINICAL TRIAL: NCT03953261
Title: Effect of Curcumin on Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID and lack of support staff 2. lack of support staff to conduct the study
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5190041
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Curcumin (Experimental)
  Interventions: Drug: Curcumin supplement
- Placebo (Placebo Comparator)
  Interventions: Drug: Curcumin supplement

INTERVENTIONS:
Drug: Curcumin supplement — Intervention is 2 grams of curcumin supplement per day

SUMMARY:
The purpose of this investigator initiated study is to determine the efficacy of curcumin on disease activity of subjects with systemic lupus erythematous. Curcumin has been found to have anti-inflammatory effects and has been found to improve disease activity in lupus patients. In addition, subjects with rheumatoid arthritis as well as osteoarthritis have also found benefit for their disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 or older
* Diagnosed with Systemic Lupus Erythematous according to the 2012 Systemic Lupus International Collaborating Clinics Classification Criteria.
* SLEDAI score of 6 or higher
* Ability to take oral medication and be willing to adhere to the study drug regimen

Exclusion Criteria:

* Inability to provide written consent for study participation
* Use of curcumin supplements within 30 days of enrollment of study
* Liver function disorders (AST/ALT > 2.5x upper limit of normal)
* Pregnancy or lactation
* Known allergic reactions to turmeric
* Subjects who are admitted for recent hospitalization within past 60 days
* Treatment with another investigational drug or other intervention within past 60 days
* Subjects with end stage renal disease on dialysis
* Subjects who lack the ability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Change in SLEDAI | 90 days
  Number of participants with change in SLEDAI by 2 points by Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No